CLINICAL TRIAL: NCT04987125
Title: Dyspnea Neuroscience Education on Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Luis Suso, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-07-15; First posted 2021-08-03 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Dyspnea
Keywords: Education; Neuroscience education
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyspnea Neuroscience education (Experimental)
  Interventions: Behavioral: Dyspnea Neuroscience education
- Usual care (Active Comparator)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Dyspnea Neuroscience education — Patients will follow an online therapeutic education course about dyspnea. Education about the cognitive and emotional aspects of dyspnea processing, with the goal of changing maladaptive cognitions and behaviors.
  The course will be group-based (5 participants). The frequency will be of 1 session per week for 4 weeks, each session will have a duration of 1 hour.
  Arms: Dyspnea Neuroscience education
Behavioral: Usual care — General health advice, physiotherapy treatment. The frequency will be of 1 session per week for 4 weeks, each session will have a duration of 1 hour.
  Arms: Usual care

SUMMARY:
The principal aim of this study was to adapt pain neuroscience education to dyspnea, Dyspnea Neuroscience Education (DNE), and measure its effect on dyspnea perception, physica l activity level, disability, quality of life and ventilatory and functional capacity through a randomized controlled trial. The secondary objectives were to evaluate its feasibility and its effect on emotional state (anxiety and depression), medical atten dance, number of exacerbations and the willingness to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of COPD by a physician or pneumologist
* Stage 1, 2 or 3 on the GOLD Classification
* GOLD Stage and FEV1 assessed by a physician in the last three months
* Access to a computer and internet

Exclusion Criteria:

* Cognitive impairment (MoCA-S score < 21)
* Depression disorder (PHQ-9 score ≥11)
* Generalized Anxiety Disorder (GAD-7 score ≥10)
* Instable comorbidities preventing physical activities
* Had a surgery in the past three months
* Had an exacerbation in the past three months
* Currently quitting tobacco
* Use of oxygenation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from Perception of Dyspnea questionnaire at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).
Change from disability questionnaire at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).
Change from Quality of Life about respiratory disease questionnaire at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).
Change from Level of Physical Activity questionnaire at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).
Change from Activity-related intensity and unpleasantness of perceived dyspnea questionnaire at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).
Change from Self-efficacy Scale for Physical Activity questionnaire at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).

SECONDARY OUTCOMES:
Change from Forced vital capacity physiological parameter at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).
Change from FEV1 physiological parameter at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).
Change from Six Minute Walk Test (Sp02% Change) physiological parameter at 4 and weeks and 6 months | Preintervention, postintervention (4 weeks) and follow-up (6 months).

IPD SHARING:
Plan to Share IPD: Undecided